CLINICAL TRIAL: NCT04480866
Title: Developing a Complete Cervical Cancer Screening Solution Based on First-void Urine Self-sampling: Improved and Quality Assured Collection of First-void Urine
Brief Title: CASUS: Improved and Quality Assured Collection of First-void Urine
Acronym: CASUS-WP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Novosanis NV (Industry); Self-screen B.V. (Unknown)
Responsible Party: Principal Investigator, Pierre Van Damme, Principal Investigator, Universiteit Antwerpen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B300201940120
Record Dates: First submitted 2020-06-02; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia; Human Papilloma Virus; HPV-Related Cervical Carcinoma; Urine
Keywords: Biomarker; First-void urine; Screening; Triage
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First-void urine collection (Other): Women self-collect three first-void urine samples (random order) at home.
  Interventions: Device: Colli-Pee® (FV5000 and Small Volumes)

INTERVENTIONS:
Device: Colli-Pee® (FV5000 and Small Volumes) — Colli-Pee® device (Novosanis, Belgium) attached to collector tubes prefilled with a non-toxic nucleic acid preservative (including an internal process control). The collector tubes differ in size to collect a total sample volume of 4, 10, and 20 mL.
  Each participant will collect three urine samples using the Colli-Pee Small Volumes 4 and 10 mL, and the Colli-Pee FV5000 (20 mL) device, in a random order.

SUMMARY:
The goal of the overall CASUS project is to develop the first fully molecular integrated cervical cancer screening approach, based on first-void urine as an easily accessible and non-invasive source of biomarkers. In contrast to current screening modalities, the CASUS approach will identify women with clinically relevant disease in need of treatment using only a single sample that can be collected at home (one-step triage).

DETAILED DESCRIPTION:
CASUS work package 1 (WP1): To accommodate for the detection of biomarkers in first-void urine, a next-generation first-void urine collection device is necessary, which includes internal process control, novel collector tubes for collection of smaller urine volumes, and integration of a non-toxic nucleic acid preservative.

Hereto, new generations of the Colli-Pee® (Novosanis) first-void urine collector allowing collection of smaller volumes (Colli-Pee Small Volumes 4 and 10 mL) next to the 'standard' Colli-Pee FV5000 (20 mL) first-void urine collector will be developed and validated. The optimal urine volume needed for detection of host and viral biomarkers, as well as optimization of the nucleic acid preservative solution by introduction of a sample/extraction validation control (non-human DNA internal control (DNA IC)) will be evaluated by measuring the concentration of human DNA, HPV DNA, and the DNA IC in all first-void urine samples using different DNA extraction protocols.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years and older
* Women with a high-risk HPV positive test result within six months prior to study enrolment.
* Giving informed consent to the research team to contact his/her general practitioner and/or gynaecologist to access details of the participants HPV test results and cervical screening history.
* Able to understand the information brochure/what the study is about.

Exclusion Criteria:

* Women that underwent hysterectomy or were treated for cervical (pre)cancer lesions within the previous six months prior to study enrolment.
* Participating in another interventional clinical study (where e.g. a medical device, drug, or vaccine is evaluated) at the same time of participating in this study. Participation in another observational or low-interventional clinical study at the same time is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Human DNA (GAPDH) | Evaluation/testing when all samples are collected [1 year]
  Comparison of human DNA (GAPDH) concentrations [cycle threshold values] between first-void urine volumes (4, 10, 20 mL) and extraction methods measured by quantitative PCR (qPCR).
Internal control DNA (IC DNA) | Evaluation/testing when all samples are collected [1 year]
  Comparison of internal control DNA (IC DNA) concentrations [cycle threshold values] between first-void urine volumes (4, 10, 20 mL) and extraction methods measured by quantitative PCR (qPCR).
Human DNA reference gene (ACTB) | Evaluation/testing when all samples are collected [1 year]
  Comparison of human DNA reference gene (ACTB) concentrations [cycle threshold values] between first-void urine volumes (4, 10, 20 mL) and extraction methods measured by quantitative methylation specific PCR (qMSP).

SECONDARY OUTCOMES:
Human DNA (Beta-globin) | Evaluation/testing when all samples are collected [1 year]
  Comparison of human DNA (Beta-globin) concentrations [cycle threshold values] between first-void urine volumes (4, 10, 20 mL) and extraction methods measured using the HPV-risk assay (Self-Screen BV).
HPV DNA (HPV16, HPV18, other high-risk HPV (HPV31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66, -67, and -68)) | Evaluation/testing when all samples are collected [1 year]
  Comparison of HPV DNA (HPV16, HPV18, other high-risk HPV (HPV31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66, -67, and -68)) positivity (+/-) and concentrations [cycle threshold values] between first-void urine volumes (4, 10, 20 mL) and extraction methods measured using the HPV-risk assay (Self-Screen BV).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, MD, PhD, Principal Investigator — Universiteit Antwerpen; Alex Vorsters, Ir, PhD, Study Chair — Universiteit Antwerpen; Severien Van Keer, PhD, Study Chair — Universiteit Antwerpen; Laura Téblick, Ir, Study Chair — Universiteit Antwerpen
Locations (1):
- Centre for the Evaluation of Vaccination (CEV) - Vaccine & Infectious Disease Institute (VAXINFECTIO) - University of Antwerp, Wilrijk, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No